CLINICAL TRIAL: NCT01057069
Title: Randomized Phase II/III Study of Individualized Neoadjuvant Chemotherapy in ' Triple Negative' Breast Tumors
Brief Title: Neo Adjuvant Chemotherapy in Triple Negative Breast Cancer
Acronym: neo-TN
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M09TNM; 2009-015238-31 (EudraCT Number)
Record Dates: First submitted 2010-01-26; First posted 2010-01-27 (Estimated); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Breast Cancer
Keywords: Neo adjuvant; Triple negative; primary tumor over 2 cm and/or positive lymphnodes
MeSH Terms: conditions — Breast Neoplasms | interventions — Carboplatin; Paclitaxel; AC protocol; Doxorubicin; Cyclophosphamide; Thiotepa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- HRD; 1x ddAC, 2x tCTC (Experimental): HRD positive tumors; irrespective of response; - a fourth course of AC followed by Peripheral Blood Progenitor Cell (PBPC) harvest and tandem intermediate-dose alkylating therapy (miniCTC, carboplatin 800 mg/m2, thiotepa 250 mg/m2, and cyclophosphamide 3000 mg/m2) with PBPC-reinfusion.
  Interventions: Drug: Doxorubicin, cyclophosphamide, carboplatin, thiotepa, cyclophosphamide
- HRD; 3x CP (Active Comparator): HRD tumors; any response to 3x ddAC; 3 courses of CP
  Interventions: Drug: Carboplatin and Paclitaxel
- non-HRD;3x CP (Active Comparator): non-HRD tumors; unfavourable response to 3x ddAC; 3 courses of Carboplatin and Paclitaxel
  Interventions: Drug: Carboplatin and Paclitaxel
- non-HRD; response; 3x ddAC (Active Comparator): non-HRD tumors; favourable response to 3x ddAC; 3 more courses of ddAC
  Interventions: Drug: Doxorubicin, cyclophosphamide
- non-HRD; response; 3x CP (Active Comparator): non-HRD tumors; favourable response to 3x ddAC; 3 courses of Carboplatin and Paclitaxel
  Interventions: Drug: Carboplatin and Paclitaxel

INTERVENTIONS:
Drug: Carboplatin and Paclitaxel — Carboplatin AUC = 6, Q 3 weeks, 3 courses Paclitaxel 80 mg/m2, weekly, 9 administrations
  Other Names: Carboplatin; Paclitaxel
  Arms: HRD; 3x CP; non-HRD; response; 3x CP; non-HRD;3x CP
Drug: Doxorubicin, cyclophosphamide — Two-weekly administrations of 600 mg/m2 cyclophosphamide and 60 mg/m2 doxorubicin PEG-filgrastim (Neulasta(r)) will be administered on the day following chemotherapy.
  Arms: non-HRD; response; 3x ddAC
Drug: Doxorubicin, cyclophosphamide, carboplatin, thiotepa, cyclophosphamide — One course of of 600 mg/m2 cyclophosphamide and 60 mg/m2 doxorubicin. PEG-filgrastim (Neulasta(r)) will be administered on the day following chemotherapy.
  This course is followed by Peripheral Blood Progenitor Cell (PBPC) harvest and tandem intermediate-dose alkylating therapy (miniCTC, carboplatin 800 mg/m2, thiotepa 250 mg/m2, and cyclophosphamide 3000 mg/m2) with PBPC-reinfusion.
  Arms: HRD; 1x ddAC, 2x tCTC

SUMMARY:
This study aims to compare the response of triple-negative breast cancer with deficient homologous recombination to intensified alkylating chemotherapy versus standard chemotherapy with dose dense AC and/or Docetaxel-Capecitabine.

DETAILED DESCRIPTION:
Homologous Recombination (HR) is a DNA repair mechanism that can repair double-strand DNA breaks. It is the only reliable repair mechanism that can repair the consequences of DNA adducts caused by bifunctional alkylating agents (such as cyclophosphamide, thiotepa or carboplatin). Alternative DNA repair mechanisms exist, but these unavoidably induce DNA mutations, deletions and chromosome aberrations, giving give rise to genetic instability. HRD may be a consequence of inactivation of the BRCA-1 or BRCA-2 genes (as in hereditary breast cancer), but it may also be caused by defects in the Fanconi anemia pathway or by amplification of the EMSY gene. HRD is present in breast cancer cells but not in healthy cells of BRCA-1 or BRCA-2 mutation carriers, and also in about half of the sporadic triple-negative breast cancers.

This phase II/III controlled multicenter trial will investigate the ability of individualized chemotherapy to improve the objective response rate of 'triple-negative' breast cancer (estrogen receptor and progesterone receptor-negative, no HER2 amplification) to preoperative (neoadjuvant) chemotherapy. It will answer the question whether intensified alkylating chemotherapy improves the response rate of tumors with a Homologous Recombination Defect (HRD) and it will gather data required for the design of a phase III study documenting the efficacy of response monitoring by contrast-enhanced MRI in TN breast cancer without HRD.

ELIGIBILITY:
Inclusion Criteria:

* Proven infiltrating breast cancer with either a primary tumor over 2 cm in size (MRI or ultrasound examination) and/or cytologically proven spread to the axillary lymph nodes.
* Patients with 'locally advanced breast cancer' are consequently eligible, including those with ipsilateral supraclavicular lymph node metastases.
* The tumor must be HER2/neu-negative (either score 0 or 1 at immunohistochemistry or negative at in situ hybridization [CISH or FISH] in case of score 2 or 3 at immunohistochemistry).
* The tumor must be Estrogen receptor (ER) -negative (< 10% nuclear staining at IHC) and Progesterone receptor (PR) -negative (< 10% nuclear staining at IHC). However, the rare tumors that are ER-negative and PR-positive will be eligible, if this pattern of hormone receptor expression can be verified in the NKI-AVL reference pathology lab.
* Age 18 to 59 years; patients older than 59 years may be included when considered 'biologically 59 years or younger' (as judged by the investigator).
* Performance status: WHO 0 or I.
* Adequate bone marrow function (W.B.C. count > 3.0 x 109/l, platelets > 100 x 109/l).
* Adequate hepatic function (ALAT, ASAT and bilirubin < 2 x upper limit of normal, or minor abnormalities of these tests judged to be of no consequence by the study coordinator).
* Adequate renal function (creatinine clearance > 60 ml/min).
* Informed consent

Exclusion Criteria:

* Previous radiation therapy or chemotherapy.
* Other malignancy except carcinoma in situ, unless the other malignancy was treated 5 or more years ago with curative intent without the use of chemotherapy or radiation therapy.
* Pregnancy or breast feeding.
* Evidence of distant metastases. Staging examinations must have included a chest roentgenogram, an ultrasound examination of the liver and an isotope bone scan. Abnormal uptake on the isotope bone scan can only be accepted if bone metastases were excluded by MRI

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 310 (Actual)
Dates: Start 2010-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
Primary endpoint (HRD tumors): Average Neoadjuvant Response Index (NRI) after intensified alkylating therapy in comparison to that after 'standard' neoadjuvant chemotherapy. Primary endpoint (non-HRD tumors): Average Neoadjuvant Response Index (NRI) | end of neo adjuvant chemotherapy

SECONDARY OUTCOMES:
Recurrence-free survival and overall survival. | every year

CONTACTS AND LOCATIONS:
Overall Officials: Sjoerd Rodenhuis, MD, Principal Investigator — NKI-AvL
Locations (14):
- Netherlands (14):
  - Medisch Centrum Alkmaar, Alkmaar
  - NKI-AVL, Amsterdam
  - OLVG, Amsterdam
  - Reinier de Graaf Groep, Delft
  - Deventer Ziekenhuis, Deventer
  - Albert Schweitzer ziekenhuis, Dordrecht
  - Ziekenhuis Gelderse Vallei, Ede
  - Kennemer Gasthuis, Haarlem
  - Atrium Medisch Centrum Parkstad, Heerlen
  - Spaarne Ziekenhuis, Hoofddorp
  - LUMC, Leiden
  - Maasstad ziekenhuis, Rotterdam
  - Medisch Centrum Haaglanden, The Hague
  - Isala Klinieken, Zwolle

REFERENCES:
- [Background] Rodenhuis S, Mandjes IAM, Wesseling J, van de Vijver MJ, Peeters MTDFV, Sonke GS, Linn SC. A simple system for grading the response of breast cancer to neoadjuvant chemotherapy. Ann Oncol. 2010 Mar;21(3):481-487. doi: 10.1093/annonc/mdp348. Epub 2009 Aug 28. PMID 19717533
- [Derived] Vliek S, Hilbers FS, van Werkhoven E, Mandjes I, Kessels R, Kleiterp S, Lips EH, Mulder L, Kayembe MT, Loo CE, Russell NS, Vrancken Peeters MTFD, Holtkamp MJ, Schot M, Baars JW, Honkoop AH, Vulink AJE, Imholz ALT, Vrijaldenhoven S, van den Berkmortel FWPJ, Meerum Terwogt JM, Schrama JG, Kuijer P, Kroep JR, van der Padt-Pruijsten A, Wesseling J, Sonke GS, Gilhuijs KGA, Jager A, Nederlof P, Linn SC. High-dose alkylating chemotherapy in BRCA-altered triple-negative breast cancer: the randomized phase III NeoTN trial. NPJ Breast Cancer. 2023 Sep 9;9(1):75. doi: 10.1038/s41523-023-00580-9. PMID 37689749
- [Derived] Miquel-Cases A, Retel VP, van Harten WH, Steuten LM. Decisions on Further Research for Predictive Biomarkers of High-Dose Alkylating Chemotherapy in Triple-Negative Breast Cancer: A Value of Information Analysis. Value Health. 2016 Jun;19(4):419-30. doi: 10.1016/j.jval.2016.01.015. Epub 2016 Apr 6. PMID 27325334
- [Derived] Miquel-Cases A, Steuten LM, Retel VP, van Harten WH. Early stage cost-effectiveness analysis of a BRCA1-like test to detect triple negative breast cancers responsive to high dose alkylating chemotherapy. Breast. 2015 Aug;24(4):397-405. doi: 10.1016/j.breast.2015.03.002. Epub 2015 Apr 28. PMID 25937263